CLINICAL TRIAL: NCT00826748
Title: Effect of Inhaled Steroids on Gene Expression in the Lungs of Healthy Smokers
Brief Title: Effect of Inhaled Steroids on Gene Expression in the Lungs - 2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 0809009975
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; inhaled steroids; gene expression; smoker's lungs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treated Smokers (Experimental): The treatment with inhaled beclomethasone will be administered to this cohort from Day 1 to Day 7 via a metered dose inhaler (QVAR 80 HFA) delivering 80 micrograms of beclomethasone per puff. QVAR will be purchased by the Department of Genetic Medicine. The dose will be 2 puffs twice a day for 7 days.
  Interventions: Drug: Beclomethasone
- Non-Treated Smokers (No Intervention): This cohort will act as control and include healthy smokers who receive no treatment.
- Non-Smokers (No Intervention): This cohort will act as control and include healthy non-smokers who receive no treatment.

INTERVENTIONS:
Drug: Beclomethasone — The treatment with inhaled beclomethasone will be administered to Group A from Day 1 to Day 7 via a metered dose inhaler (QVAR 80 HFA) delivering 80 micrograms of beclomethasone per puff. QVAR will be purchased by the Department of Genetic Medicine. The dose will be 2 puffs twice a day for 7 days
  Other Names: QVAR 80 HFA
  Arms: Treated Smokers

SUMMARY:
The purpose of this study is to assess the effect of inhaled beclomethasone (an inhaled corticosteroid) on the pattern of the lung airway epithelium and alveolar macrophages gene expression of healthy smokers. We hypothesize that the administration of beclomethasone will result in reversibility of some of the airway epithelium and alveolar macrophage gene expression changes induced by cigarette smoking.

DETAILED DESCRIPTION:
The study will involve healthy smokers and non smokers enrolled in IRB approved protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy". They will be invited to participate in this protocol only if they meet the additional inclusion/exclusion criteria of this protocol (see inclusion/exclusion criteria, section A6). The Principal Investigator, Ann E. Tilley, MD or authorized representative will obtain consent from individuals for this study. Once enrolled, smokers will be randomized to either the treated smoker group [320 micrograms (mcg) of beclomethasone; 2 puffs twice a day (each puff delivers 80 mcg) for 7 days] or non-treated group. Beclomethasone is available as a metered dose inhaler [QVAR(TEVA Pharmaceuticals)] delivering 80 micrograms (mcg) of beclomethasone per one puff. We will be using QVAR HFA (TEVA Pharmaceuticals), which delivers 80 mcg per puff. QVAR will be purchased by the Department of Genetic Medicine. It will be dispensed as appropriate to each research subject recruited in the trial at the Department of Genetic Medicine at 1305 York Ave YAB-13th floor, New York, NY 10021 (a facility of Weill Medical College). It will be stored at The Arthur & Rochelle Belfer Gene Therapy Core Facility located at 515 E. 71st St., S901, New York, NY 10021 under the supervision of Stephen Kaminksy, PhD, Co-Director of the GMP (Good Manufacturing Practice). Each study individual will receive 1 package of the study medication which consists of 1 canister of QVAR 80 MDI (metered dose inhaler). Non-smokers, defined as individuals who have never smoked, will act as control like the Non-Treated Smoker group and receive no treatment. For all subjects, the screening, baseline bronchoscopy, and the bronchoscopies on Days 7±3 and 14±3 tests will be performed as part of IRB approved protocol #0005004439. No additional bronchoscopies will be performed under the current protocol.

ELIGIBILITY:
Inclusion Criteria:

All Smokers (Treated and Non-Treated)

* All study individual should be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"
* All study subjects should be able to provide informed consent
* Current smokers with 15-to 40 pack-year history
* All study individuals should be healthy as per protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"

Non-Smokers

* All study individual should be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"
* All study subjects should be able to provide informed consent
* All study individual should be healthy as per protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"

Exclusion Criteria:

All Smokers

* Smokers intending to quit smoking in the next 14 days.
* Individuals already receiving any lung related inhalers
* Females who are pregnant or nursing

Non-Smokers

Exclusion Criteria:

* Non-smokers who intend to start smoking in the next 14 days
* Individuals already receiving any lung related inhalers
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 subjects underwent informed consent and enrolled into the study. 2 smoker subjects screen-failed (recent illicit drug use history of myocardial infarction). These individuals were dropped from the study prior to randomization, therefore only 22 individuals were assigned into one of the three study groups.
Groups:
- Treated Smokers: The treatment with inhaled beclomethasone will be administered to Treated Smokers from Day 1 to Day 7 via a metered dose inhaler (QVAR 80 HFA) delivering 80 micrograms of beclomethasone per puff. QVAR will be purchased by the Department of Genetic Medicine. The dose will be 2 puffs twice a day for 7 days.
- Non-Treated Smokers: Non-Treated Smokers will act as control and include healthy smokers who receive no treatment.
- Non-Smokers: Non-Smokers will act as control and include healthy non-smokers who receive no treatment.
Period: Overall Study
Arm/Group | Treated Smokers | Non-Treated Smokers | Non-Smokers
Started | 6 | 4 | 12
Completed | 6 | 4 | 8
Not Completed | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Samples Did Not pass QC | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The subjects included in this group underwent the screening visit and were determined eligible to undergo the baseline assessments and sample collection procedure.
Groups:
- Non-Treated Smokers: Non-Treated Smokers will act as a control and includes healthy smokers who received no treatment.
- Non-smokers: Non-Smokers will act as a control and includes healthy non-smokers who received no treatment.
- Total: Total of all reporting groups
Arm/Group | Treated Smokers | Non-Treated Smokers | Non-smokers | Total
Number analyzed (Participants) | 6 | 4 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 12 | 22
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 7 | 8
  Male | 6 | 3 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With A Significant Change in Gene Expression in the Airway Epithelium and Alveolar Macrophages at Days 7 and 14
Description: The primary study endpoint is a change in the gene expression in the airway epithelium or alveolar macrophages of healthy smokers following treatment with beclomethasone. Airway epithelium and alveolar macrophages are processed to yield high quality RNA. Complementary DNA (cDNA) is transcribed from the RNA in vitro and the product is hybridized onto gene microarray chips. The chip is then scanned and the image analyzed using the Affymetrix Microarray suite version 5 (MAS5) algorithm. Using GeneSpring software the data is normalized and differential expression is determined by fold change (up or down regulation) of the individual genes by comparing the geometric mean expression value from the airway epithelium and alveolar macrophages obtained from Day 7 and Day 14 following initiation of therapy to baseline values.
Time Frame: Analysis will be done on samples collected on Day 7 and Day 14 following initiation of therapy compared to baseline values obtained on the day prior to initiation of treatment.
Population: Subjects underwent bronchoscopy procedure at 7 and 14 days after baseline to collect samples including small airway epithelium and alveolar macrophages.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Smokers: Non-Smokers will act as control and include healthy non-smokers who receive no treatment. Two subjects withdrew consent prior to the Day 7 timepoint, therefore only 10 subjects have data available past Day 7.
Arm/Group | Treated Smokers | Non-Treated Smokers | Non-Smokers
Number analyzed (Participants) | 6 | 4 | 10
Participants
  Small Airway Epithelium | 0 | NA — No analysis was performed for this group since: 1. There was no effect observed in the intervention group (Treated Smokers) and 2. Not enough subjects had samples collected for all timepoints obviating a meaningful analysis. | NA — No analysis was performed for this group since: 1. There was no effect observed in the intervention group (Treated Smokers) and 2. Not enough subjects had samples collected for all timepoints obviating a meaningful analysis
  Alveolar Macrophages | 0 | NA — No analysis was performed for this group since: 1. There was no effect observed in the intervention group (Treated Smokers) and 2. Not enough subjects had samples collected for all timepoints obviating a meaningful analysis. | NA — No analysis was performed for this group since: 1. There was no effect observed in the intervention group (Treated Smokers) and 2. Not enough subjects had samples collected for all timepoints obviating a meaningful analysis.

ADVERSE EVENTS:
Groups:
- Treated Smokers: Treated Smokers will be administered with 320 micrograms (mcg) of beclomethasone daily from Day 1 to Day 7 via a metered dose inhaler (QVAR 80 HFA) delivering 80 micrograms of beclomethasone per puff. The dose will be 2 puffs twice a day for 7 days.
Arm/Group | Treated Smokers | Non-Treated Smokers | Non-smokers
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/12
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/12

LIMITATIONS AND CAVEATS:
The study could not completed as designed due to a lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes